CLINICAL TRIAL: NCT00323063
Title: Randomized Phase II Trial of Gemcitabine and Imatinib Mesylate Versus Gemcitabine Alone in Patients With Previously Treated Locally Advanced or Metastatic Breast Cancer
Brief Title: Gemcitabine +/- Imatinib Mesylate, Patients w/Previously Treated Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis Pharmaceuticals (Industry); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Deborah Toppmeyer, MD, Chief, Division of Medical Oncology, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0220060081; P30CA072720 (NIH); CDR0000539445 (Other: NIH); 0220060081 (Other: IRB Number); NJ1105 (Other: CINJOG number); NCI-2012-00520 (Other: NCI); 040504 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Gemcitabine; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Gemcitabine Hydrochloride) (Active Comparator): Patients receive gemcitabine hydrochloride IV on days 3 and 10.
  Interventions: Drug: gemcitabine hydrochloride
- Arm II (Gemcitabine Hydrochloride + Imatinib) (Experimental): Patients receive gemcitabine hydrochloride IV on days 3 and 10 and oral imatinib mesylate once daily on days 1-5 and 8-12.
  Interventions: Drug: gemcitabine hydrochloride; Drug: imatinib mesylate

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
Drug: imatinib mesylate — Given orally
  Arms: Arm II (Gemcitabine Hydrochloride + Imatinib)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine together with imatinib mesylate may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying gemcitabine and imatinib mesylate to see how well they work compared to gemcitabine alone in treating patients with previously treated locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare time to progression in patients with previously treated locally advanced or metastatic breast cancer treated with gemcitabine hydrochloride with vs without imatinib mesylate.

Secondary

* Compare the efficacy of these regimens in these patients.
* Compare the overall survival of patients treated with these regimens.
* Compare the safety and tolerability of these regimens in these patients.

OUTLINE: This is a multicenter, open-label, randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV on days 3 and 10.
* Arm II: Patients receive gemcitabine hydrochloride IV on days 3 and 10 and oral imatinib mesylate once daily on days 1-5 and 8-12.

In both arms, treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Locally advanced or metastatic disease
  * Disease progression after at least 1 prior chemotherapy regimen for metastatic disease

    * No more than 2 prior chemotherapy regimens for metastatic disease (prior neoadjuvant or adjuvant treatment will not be included in determining the number of prior chemotherapy regimens)
* Measurable disease
* No known symptomatic or untreated brain metastases or carcinomatous meningitis

  * Previously treated and clinically stable brain metastases allowed provided patient has been off steroids for > 7 days
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* Able to swallow oral medication
* No coexisting medical condition that would preclude study compliance
* No uncontrolled illness, including any of the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia requiring therapy
  * Myocardial infarction within the past 6 months
  * Active infection
* No New York Heart Association class III-IV cardiac disease
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to gemcitabine hydrochloride and/or imatinib mesylate
* No other primary malignancies within the past 5 years except for carcinoma in situ of the cervix or nonmelanoma skin cancer
* No known chronic liver disease (i.e., chronic active hepatitis or cirrhosis)
* No known HIV infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* More than 2 weeks since prior surgery
* At least 2 weeks since prior hormonal therapy
* At least 2 weeks since prior trastuzumab (Herceptin®)
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* At least 3 weeks since prior anti-vascular endothelial growth factor therapy
* More than 28 days since prior investigational agents
* At least 3 weeks since prior radiotherapy

  * Must have evidence of ≥ 1 measurable target lesion outside the irradiated fields OR radiologically confirmed disease progression within the irradiated fields after completion of radiotherapy
* No prior imatinib mesylate for metastatic disease
* No prior gemcitabine hydrochloride for metastatic disease
* More than 6 months since prior adjuvant gemcitabine hydrochloride
* No other concurrent investigational or commercial agents
* No concurrent therapeutic anticoagulation with warfarin (e.g., Coumadin® or Coumadine®)

  * Concurrent heparin or low-molecular weight heparin (e.g., Lovenox®) for therapeutic anticoagulation allowed
  * Concurrent prophylactic warfarin therapy (e.g., mini-dose Coumadin® ≤ 1 mg daily) to maintain catheter patency allowed
* No concurrent routine chronic systemic corticosteroids
* No concurrent medications that would preclude study compliance

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2011-04-15 (Actual); Study Completion 2016-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah R. Toppmeyer, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (9):
- United States (9):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Rutgers Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Mountainside Hospital, Montclair, New Jersey
  - Jersey Shore Cancer Center at Jersey Shore University Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - NJ Medical School, Newark, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was opened to accural on 5/1/2006 and was closed to accrual on 4/15/2011 due to slow accrual. Subjects were recruited through the Cancer Institute of New Jersey Oncology Group. We are reporting results on 49 eligible patients. One was not eligible for participation.
Groups:
- Gemcitabine Hydrochloride: Patients receive gemcitabine hydrochloride 1250 mg/m2 intravenously on days 3 and 10.
  gemcitabine hydrochloride: Given IV
- Gemcitabine Hydrochloride + Imatinib: Patients receive gemcitabine hydrochloride 1250 mg/m2 intravenously on days 3 and 10 and oral imatinib mesylate 400 mg orally once daily on days 1-5 and 8-12.
  gemcitabine hydrochloride: Given IV
  imatinib mesylate: Given orally
Period: Overall Study
Arm/Group | Gemcitabine Hydrochloride | Gemcitabine Hydrochloride + Imatinib
Started | 26 | 23
Completed | 24 | 23
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — brain mets discovered prior to treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study was prematurely closed due to slow accrual.
Groups:
- Arm I: Patients receive gemcitabine hydrochloride 1250 mg/m2 intravenously on days 3 and 10.
  gemcitabine hydrochloride: Given IV
- Arm II: Patients receive gemcitabine hydrochloride 1250 mg/m2 intravenously on days 3 and 10 and oral imatinib mesylate 400 mg orally once daily on days 1-5 and 8-12.
  gemcitabine hydrochloride: Given IV
  imatinib mesylate: Given orally
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 11 | 10 | 21
Age, Continuous [Median (Full Range); unit: years] | 60.7 [39 to 78] | 62.4 [45 to 81] | 61.5 [39 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 24 | 22 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 17 | 16 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 23 | 49

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Sample size of 40 patients per group was needed to detect an 8 month increase in time to progression with the combination (80% power, alpha =.05, 2-sided).
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine Hydrochloride + Imatinib)
Number analyzed (Participants) | 26 | 23
months | 2 [1 to 5] | 2.5 [1 to 5]
Statistical Analysis 1: Comparison: Arm I (Gemcitabine Hydrochloride) vs Arm II (Gemcitabine Hydrochloride + Imatinib); Test type: Other; p = 0.3, Log Rank

2. Secondary Outcome: Response Rate (Complete and Partial Response)
Description: Overall response rate was evaluated every 2 cycles (six weeks) for both groups using international criteria by the Response Evaluation Criteria in Solid Tumors (RECISTv1.0) for target lesions and were assessed by CT or MRI. Response rates were defined as complete response (CR), disappearance of all target lesions; partial response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Overall response(OR) defined as OR=CR + PR
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine Hydrochloride + Imatinib)
Number analyzed (Participants) | 26 | 23
percentage of participants | 9.1 [1.6 to 30.6] | 9.1 [1.6 to 30.6]

3. Secondary Outcome: Overall Survival
Time Frame: 5 years
Population: This study was prematurely closed so overall survival was not analyzed.
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine Hydrochloride + Imatinib)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Arm I (Gemcitabine Hydrochloride): Patients receive gemcitabine hydrochloride 1250 mg/m2 intravenously on days 3 and 10.
  gemcitabine hydrochloride: Given IV
- Arm II (Gemcitabine Hydrochloride + Imatinib): Patients receive gemcitabine hydrochloride 1250 mg/m2 intravenously on days 3 and 10 and oral imatinib mesylate 400 mg orally once daily on days 1-5 and 8-12.
  gemcitabine hydrochloride: Given IV
  imatinib mesylate: Given orally
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine Hydrochloride + Imatinib)
All-Cause Mortality (participants affected / at risk) | 0/26 | 2/23
Serious Adverse Events (participants affected / at risk) | 5/26 | 6/23
Other Adverse Events (participants affected / at risk) | 26/26 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Gemcitabine Hydrochloride) (N=26) | Arm II (Gemcitabine Hydrochloride + Imatinib) (N=23)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neutrophils decreased (Investigations) | 0 (0) | 1 (1)
Anemia (Investigations) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Gemcitabine Hydrochloride) (N=26) | Arm II (Gemcitabine Hydrochloride + Imatinib) (N=23)
alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Alanine aminotransferase (Investigations) | 4 (5) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Fatigue (General disorders) | 10 (16) | 4 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 13 (31) | 8 (40)
White blood cell decreased (Investigations) | 14 (30) | 7 (39)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 20 (45) | 10 (57)
Platelet count decreased (Investigations) | 7 (16) | 5 (20)
Vomiting (Gastrointestinal disorders) | 5 (6) | 3 (11)
Nausea (Gastrointestinal disorders) | 9 (12) | 5 (17)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (5)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1)
Aspartate aminoransferase elevated (Investigations) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 5 (5) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was underpowered to draw any conclusion regarding a difference in TTP between the two groups at the time is was prematurely closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Informed Consent Form (2009-12-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT00323063/ICF_000.pdf